CLINICAL TRIAL: NCT06704776
Title: The Medially Pedicled Infrapatellar Fat Pad (IPFP) ﬂap in Total Knee Arthroplasty (TKA)
Brief Title: The Medially Pedicled IPFP ﬂap in TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Fang, Deputy chief physician, First Affiliated Hospital of Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU|2023]376
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-01

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis (OA)
Keywords: Total knee arthroplasty; IPFP; Knee osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The trial employs a random allocation method. A randomization table will be generated using SPSS 26.0 software. Treatment groups will be selected based on patients' random numbers, ensuring that this clinical institution stratifies the subjects into an "The medially pedicled IPFP flap" group and a "Complete IPFP removal" group at a 1:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers, outcome assessors and statisticians will be blinded to the group assignments and will not be involved in the trial operations. The patients will also be blinded to the group assignments. Due to the impossibility of blinding the surgeons, they will not be involved in any outcome assessments. Allocation results will be placed in sealed envelopes before the surgery. The envelopes will be opened prior to surgery after the administration of general anaesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "The medially pedicled IPFP flap" group (Experimental): In the "The medially pedicled IPFP flap" group, the IPFP was exposed and separated, and the lateral side was left intact and the medial side was tipped to form a complete medially tipped IPFP flap, and the IPFP flap was clipped and draped over the medial side to avoid interference of the IPFP with the operative field. After successful implantation of the prosthesis, the IPFP was fixed with in situ sutures.
  Interventions: Procedure: "The medially pedicled IPFP flap" group
- "Complete IPFP removal" group (Active Comparator): In the "Complete IPFP removal" group, the entire IPFP was resected from below the patellar tendon prior to femoral preparation.
  Interventions: Procedure: "Complete IPFP removal" group

INTERVENTIONS:
Procedure: "The medially pedicled IPFP flap" group — In the "The medially pedicled IPFP flap" group, the IPFP was exposed and separated, and the lateral side was left intact and the medial side was tipped to form a complete medially tipped IPFP flap, and the IPFP flap was clipped and draped over the medial side to avoid interference of the IPFP with the operative field. After successful implantation of the prosthesis, the IPFP was fixed with in situ sutures.
  Arms: "The medially pedicled IPFP flap" group
Procedure: "Complete IPFP removal" group — The entire IPFP was resected from below the patellar tendon prior to femoral preparation.
  Arms: "Complete IPFP removal" group

SUMMARY:
This is a single-center prospective cohort study in which patients were evaluated by inclusion and exclusion criteria before total knee arthroplasty (TKA). Eligible patients will be included in this study after signing the informed consent form. These patients will be randomly assigned to an experimental group ("The medially pedicled IPFP flap" group) and a control group ("complete IPFP removal" group). Patients were unaware of their grouping and were operated on by the same experienced surgeon. The surgical steps are identical except for the different management of the IPFP. Assessment of knee function will be performed at baseline, preoperatively, and during the 3 weeks, 3 months, 6 months and 12 months postoperative follow-up periods to evaluate the patients' prognostic outcomes. The study will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines for reporting parallel group randomised trials. Ethical approval will be obtained from each institution. Written informed consent will be obtained from all participants to ensure their voluntary participation and understanding of the study.

DETAILED DESCRIPTION:
This is a single-center prospective cohort study in which patients were evaluated by inclusion and exclusion criteria before total knee arthroplasty (TKA). This study aims to recruit 200 patients across a single centre over 1 year. Eligible patients will be included in this study after signing the informed consent form. Before TKA, the patients will be randomly assigned to either an experimental group ("The medially pedicled IPFP flap" group) or a control group ("complete IPFP removal" group) and administered different management of the IPFP during surgery. Assessment of knee function will be performed at baseline, preoperatively, and during the 3 weeks, 3 months, 6 months and 12 months postoperative follow-up periods to evaluate the patients' prognostic outcomes. The primary outcomes are the intraoperative bleeding, the visual analogue scale (VAS) score and Knee Injury and Osteoarthritis Outcome Score (KOOS). Secondary outcomes include American Knee Society Knee Score (KSS), Insall-Salvati Ratio (ISR) and knee joint range of motion (ROM). All patients voluntarily participated in the study and signed informed consent. During the treatment period, all prospective patients underwent clinical evaluation at the end of total knee arthroplasty and 3 weeks, 3 months, 6 months and 12 months later, aimed at comparing the postoperative pain and inflammatory response between "The medially pedicled IPFP flap" group and "complete IPFP removal" group, to explore the optimal perioperative analgesic modality for TKA. Statistical analyses utilizing regression models and survival analysis will be conducted to assess the relationships between the management of the IPFP and postoperative efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of primary KOA confirmed by imaging (KL classification >=2)
2. Surgeon's opinion of eligibility for primary unilateral total knee arthroplasty (TKA) based on standard evaluation procedures
3. Age: 40-80 years, male and female
4. The patient volunteers to participate in the study by signing an informed consent form for either the 'medial attachment tipped IPFP flap' or the 'complete resection of the IPFP' approach.
5. Patients understand the study requirements and are willing to co-operate with the study instructions.

Exclusion Criteria:

1. History of previous surgical knee surgery or surgical knee infection
2. Patients with a diagnosis other than osteoarthritis (including rheumatoid arthritis, traumatic arthritis, septic arthritis and haemophilic arthritis)
3. Severe osteoarthritis (including flexion contracture >30 or inversion/eversion deformity >30, and use of non-traditional restrictive joint prosthesis due to complex joint pathology)
4. presence of neuromuscular dysfunction on the operated side
5. The surgeon considers that other surgical modalities (UKA, HTO, revision surgery) are appropriate for treatment according to the standard assessment process
6. The patient decides to use other partial IPFP preservation options
7. Poor overall health conditions, including but not limited to a glycated haemoglobin level exceeding 12%, blood pressure exceeding 170/110 mmHg, myocardial infarction, stroke, transient ischaemic attack, acute congestive heart failure, or any acute coronary events within the past 6 months, severe hepatic or renal dysfunction, pregnancy, lactation and possible or planned pregnancy, history of psoriatic arthritis, lupus or cancer and psychiatric, cognitive and/or neurological disorders
8. Concurrent participation in a clinical trial other than this trial
9. Patients who, in the judgement of the investigator, no longer meet the criteria for the study due to adherence issues

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-01-29 (Estimated); Study Completion 2026-01-29 (Estimated)

PRIMARY OUTCOMES:
Intraoperative bleeding | 4 days postoperatively
  Intraoperative bleeding will be estimated by subtracting the preoperative hemoglobin level from the hemoglobin level measured 24 hours postoperatively and the preoperative hemoglobin level from the hemoglobin level measured 4 days postoperatively.
Postoperative visual analogue scale (VAS) scores at 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA | 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  VAS scores are the most commonly used indicator for assessing the intensity of patient pain. The scale ranges from "0" to "10", where "0" indicates no pain and "10" represents the most severe pain that is unbearable. Patients will rate their pain based on subjective perceptions. In this trial, VAS scores will be recorded once before TKA. The VAS scores will be assessed separately for the resting and flexion states. If the patient's hospitalization period is shorter than 72 hours, the VAS score at discharge will be recorded instead of that at 72 hours. The results will be used to evaluate whether "IPFP flap with pedicle medial attachment " can reduce pain after TKA.
Total Knee Injury and Osteoarthritis Outcome Score (KOOS) at 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA | 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  The KOOS is a patient-reported questionnaire for the knee that includes 42 items in five separately analysed subscales for pain, other symptoms, function in daily living, sport and recreational function and knee-related quality of life.Scores from 0-100 will be converted to the appropriate scale, with 0 representing severe knee problems and 100 representing no problems.The KOOS has been validated for use in TKA and has been shown to be a valid and reliable assessment measure.
Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales for pain at 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA | 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  The KOOS is a patient-reported questionnaire for the knee that includes 42 items in five separately analysed subscales for pain, other symptoms, function in daily living, sport and recreational function and knee-related quality of life.Scores from 0-100 will be converted to the appropriate scale, with 0 representing severe knee problems and 100 representing no problems.The KOOS has been validated for use in TKA and has been shown to be a valid and reliable assessment measure.
Total morphine consumption during hospitalization | through study completion, an average of 6 months
  It will be converted to total morphine equivalents and will include both the postoperative routine pain management regimen and extra analgesia.

SECONDARY OUTCOMES:
American Knee Society Knee Score (KSS) | 1-5 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  The KSS score is a comprehensive scoring system consisting of two components: the knee score and the functional score. The knee score includes ratings of pain, mobility, and stability, with a subtraction for knee deformity. The functional score includes ratings of walking ability and ability to walk up and down stairs. Both scores range from 0-100, with higher scores being associated with better function.The KSS has been used to document and report postoperative functional outcomes of TKA worldwide.
Insall-Salvati Ratio (ISR) | 3 weeks, 3 months, 6 months and 12 months after TKA
  The Insall-Salvati Ratio (ISR) is used to assess changes in patellar tendon length at baseline and at 3 weeks, 3 months, 6 months, and 12 months postoperatively. Experienced radiographers will use standardised radiography to take lateral photographs of the knee flexed at approximately 30° The numerator of the ISR is the length of the patellar tendon (the distance from the inferior aspect of the patella to the superior aspect of the tibial tuberosity on the lateral radiograph) The denominator of the ISR is the longest dimension of the patella on the lateral radiograph.
Range of motion (ROM) | 3 weeks, 3 months, 6 months and 12 months after TKA
  The range of motion (ROM) will be measured with a protractor thrice daily at 6-hour intervals, and the best value on each day will be used in the analysis. The range of motion (ROM) is from 0 to 180 degrees. The larger the angle, the more satisfactory the recovery of joint function.

OTHER OUTCOMES:
Complete blood count | 1 day, 4 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  A complete blood count (CBC) can reflect the patient's postoperative inflammatory status. It measures various components of the blood, including white blood cells, red blood cells, and platelets, which can indicate the presence of inflammation or infection. An elevated white blood cell count, for example, is often associated with an inflammatory response.
C-reactive protein (CRP) | 1 day, 4 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  C-reactive protein (CRP) can reflect the patient's postoperative inflammatory status.
Erythrocyte sedimentation rate (ESR) | 1 day, 4 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  Erythrocyte sedimentation rate (ESR) can reflect the patient's postoperative inflammatory status.
Interleukin-6 (IL-6) | 1 day, 4 days, 3 weeks, 3 months, 6 months and 12 months after TKA
  Interleukin-6 (IL-6) can reflect the patient's postoperative inflammatory status.
Massachusetts Medical Imaging (MRI) | 3 months and 12 months after TKA
  MRI can be used to assess the position of the prosthesis and the status of the surrounding soft tissues after TKA.
Age | through study completion, an average of 1 year
  Age in years will be obtained from the electronic medical records system.
Sex | through study completion, an average of 1 year
  Sex (male or female) will be obtained from the electronic medical records system.
Operative site | through study completion, an average of 1 year
  Operative site (left or right) will be obtained from the electronic medical records system.
BMI | through study completion, an average of 1 year
  Weight (kg) and height (m) will be combined to report BMI in kg/m^2, which will be obtained from the electronic medical records system. This information will be collected by the same evaluator and used to calculate the age-corrected Charlson Comorbidity Index (aCCI), baseline ROM, HSS score and VAS score for these patients.
Time to discharge | through study completion, an average of 1 year
  Time to discharge will be sourced from the electronic medical records system and used to evaluate the impacts of PSIA and PLIA on the surgical process and postoperative recovery.
Incidence of Adverse events (AEs) | through study completion, an average of 1 year
  Adverse events (AEs) are adverse medical events that occur in clinical trial subjects after receiving treatment. In this study, total AEs will be mainly categorized into local AEs and systemic AEs. Local AEs include but are not limited to prolonged wound drainage (wound drainage persists on postoperative day 3, and the drainage area of the wound dressing is greater than 2×2 cm , poor wound healing and prosthetic joint infection. Systemic AEs include but are not limited to deep vein thrombosis events, systemic infection and serious adverse events such as pulmonary embolism and death.

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Zhang, MD, Study Director — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University,, Fuzhou, Fujian, China